CLINICAL TRIAL: NCT07043621
Title: Scalp Block Before Incision or Before Emergence in Craniotomy: A Randomized Controlled Evaluation of Effectiveness and Recovery Quality Via QoR-40
Brief Title: When to Block? Timing of Scalp Block in Craniotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Muhammed Halit Tekeci, MD, Anesthesiology and Reanimation Specialist, M.D., Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-43012747-050.04-474853246
Record Dates: First submitted 2025-06-18; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Scalp Block; Regional Anesthesia; Craniotomy Surgery; QoR-40
Keywords: Scalp Block; Craniotomy surgery; analgesia; postoperative pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A total of 60 patients undergoing elective craniotomy will be randomly assigned to one of two parallel groups (n=30 per group). Group 1 will receive a preoperative scalp block, while Group 2 will receive a postoperative scalp block. A blinded investigator will monitor intraoperative hemodynamic parameters and assess both intraoperative and postoperative opioid and analgesic consumption. Postoperatively, all patients will complete the validated Quality of Recovery-40 (QoR-40) questionnaire to evaluate recovery outcomes. The study aims to compare the effect of scalp block timing on postoperative recovery and analgesic requirements.
Who Masked: Participant, Outcomes Assessor
Masking Description: A blinded investigator will monitor intraoperative hemodynamics, evaluate opioid/analgesic use, and assess postoperative recovery using the QoR-40 questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Scalp Block Group (Active Comparator): Patients in this group will receive a scalp block with 0.25% bupivacaine (20 mL) administered under ultrasound guidance after the induction of general anesthesia but prior to head pinning
  Interventions: Procedure: Early Scalp Block Group
- Postoperative Scalp Block Group (Active Comparator): Patients in this group will receive a scalp block with 0.25% bupivacaine (20 mL) administered under ultrasound guidance at the end of surgery, before emergence from anesthesia.
  Interventions: Procedure: Late Scalp Block Group

INTERVENTIONS:
Procedure: Early Scalp Block Group — Following induction of general anesthesia and prior to head pinning (Mayfield clamp placement), a scalp block was performed under aseptic conditions using 20 mL of 0.25% bupivacaine.
  The block targeted six sensory nerves that innervate the scalp: Supraorbital nerve, Supratrochlear nerve, Auriculotemporal nerve ,Zygomaticotemporal nerve, Greater occipital nerve, Lesser occipital nerve.
  Each nerve was infiltrated subcutaneously at its anatomical location using a 25-gauge needle, with the total volume distributed evenly or proportionally across the injection sites.
  Other Names: Pre-pinning Scalp Block Group
  Arms: Early Scalp Block Group
Procedure: Late Scalp Block Group — In the pre-emergence group, the scalp block was performed at the end of surgery but before emergence from general anesthesia, while the patient was still under deep anesthesia.
  Under strict aseptic conditions, 20 mL of 0.25% bupivacaine was administered to block the following six sensory nerves innervating the scalp: Supraorbital nerve, Supratrochlear nerve, Auriculotemporal nerve, Zygomaticotemporal nerve, Greater occipital nerve, Lesser occipital nerve.
  The local anesthetic was injected subcutaneously at the anatomical landmarks of each nerve using a 25-gauge needle. The total volume was distributed evenly or proportionally depending on the area. No additional surgical stimulation occurred after the block, and extubation followed routine emergence from anesthesia.
  Other Names: Pre-emergence Scalp Block Group
  Arms: Postoperative Scalp Block Group

SUMMARY:
This study aims to evaluate the effect of scalp block timing-whether administered preoperatively or postoperatively-on postoperative recovery quality in patients undergoing craniotomy. The recovery quality will be assessed using the validated Quality of Recovery-40 (QoR-40) questionnaire. A total of 60 patients, aged 18-80 years, classified as ASA I-III and with a Glasgow Coma Scale (GCS) score of 15 upon admission to the recovery unit, will be enrolled. The primary outcome is the QoR-40 score. Secondary outcomes include hemodynamic changes and pain intensity measured by the Visual Analog Scale (VAS).

DETAILED DESCRIPTION:
Craniotomy is a surgical procedure involving the opening of the skull to access the brain. Awakening patients after craniotomy must be performed gradually to maintain hemodynamic stability. During the procedure, injury to soft tissues and muscles can lead to somatic pain, which may cause hypertension and tachycardia, potentially increasing intracranial pressure and resulting in cerebral edema or hematoma. Therefore, effective postoperative pain management and hemodynamic stability are crucial in neurosurgical patients.

Post-craniotomy pain control methods include opioids, non-steroidal anti-inflammatory drugs (NSAIDs), local anesthetic infiltration at the incision site, and scalp block. However, prolonged opioid use is not recommended due to the risk of dependence and negative cognitive effects. Scalp block has been shown to be effective in controlling post-craniotomy pain and offers prolonged analgesia.

The Quality of Recovery-40 (QoR-40) questionnaire, developed by P.S. Myles, is a validated tool used to assess postoperative recovery. It is a five-point Likert-type scale consisting of 40 items, divided into five subscales: emotional state (9 items), physical comfort (12 items), psychological support (7 items), physical independence (5 items), and pain (7 items). Total scores range from 40 to 200, with higher scores indicating better recovery.

While the efficacy of scalp block in post-craniotomy pain control is well established, limited data exist regarding the influence of timing of block administration on recovery quality. This study aims to compare the effects of preoperative versus postoperative scalp block on recovery, using the QoR-40 questionnaire.

A total of 60 patients undergoing craniotomy at Sakarya University Training and Research Hospital will be included. Eligibility criteria include patients aged 18-80 years, classified as ASA I-III, and with a postoperative GCS of 15. Exclusion criteria include chronic preoperative use of analgesics, GCS <15, known allergy to local anesthetics or opioids used in scalp block or patient-controlled analgesia.

The primary outcome is the QoR-40 score. Secondary outcomes include intraoperative and postoperative hemodynamic parameters and postoperative pain scores measured with the Visual Analog Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years.
* Scheduled for craniotomy under general anesthesia.
* ASA physical status classification I to III.
* Glasgow Coma Scale (GCS) score of 15 at the time of emergence from anesthesia.
* Provide informed consent to participate in the study.

Exclusion Criteria:

* Chronic use of analgesic medications prior to surgery.
* Glasgow Coma Scale (GCS) score below 15 postoperatively.
* Allergy or hypersensitivity to local anesthetics or opioids used in the study.
* Contraindications for scalp block or patient-controlled analgesia.
* Patients with severe hepatic, renal, or cardiac dysfunction.
* Patients unable to comprehend or complete the QoR-40 questionnaire.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery Score | The observation period extended from the beginning of surgery until 24 hours postoperatively.
  Patient recovery will be assessed using the validated Turkish version of the QoR-40 (Quality of Recovery-40) questionnaire, a 40-item Likert-type scale covering five domains: emotional state, physical comfort, psychological support, physical independence, and pain. The total score ranges from 40 (poor recovery) to 200 (excellent recovery).

SECONDARY OUTCOMES:
Perioperative Hemodynamic Changes | Intraoperative (Hemodynamic parameters were monitored from the beginning to the end of surgery.)
  Heart rate will be recorded at the following time points:
  Baseline (before anesthesia induction)
  Before head pinning
  1 minute after head pinning
  30 minutes after surgical incision
  60 minutes after surgical incision
  90 minutes after surgical incision
  Before extubation
  At the 5th minute after extubation
  These measurements will be used to evaluate intraoperative hemodynamic stability between study groups.
Perioperative Hemodynamic Changes | Intraoperative (Hemodynamic parameters were monitored from the beginning to the end of surgery.)
  mean arterial pressure (MAP) will be recorded at the following time points:
  Baseline (before anesthesia induction)
  Before head pinning
  1 minute after head pinning
  30 minutes after surgical incision
  60 minutes after surgical incision
  90 minutes after surgical incision
  Before extubation
  At the 5th minute after extubation
  These measurements will be used to evaluate intraoperative hemodynamic stability between study groups.
Intraoperative and Postoperative Opioid Consumption | Total opioid consumption will be recorded intraoperatively and within the first 24 hours postoperatively.
  From induction to 24 hours postoperatively
Postoperative Pain Scores | 10 minutes, 2 hours, 6 hours, and 24 hours postoperatively
  Pain will be assessed using a 10-point Visual Analog Scale (VAS), where 0 indicates no pain and 10 indicates the worst imaginable pain.

OTHER OUTCOMES:
Adverse effects | Postoperative 24 hours
  Any adverse effects related to anesthetic and analgesic procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University Training and Research Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided